CLINICAL TRIAL: NCT01746667
Title: Virtual Reality Exposure Therapy Versus Exposure in Vivo for Social Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05510207
Record Dates: First submitted 2012-11-19; First posted 2012-12-11 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Social Anxiety Disorder; Social Phobia
Keywords: Social Anxiety Disorder; Social Phobia; Virtual Reality; Exposure
MeSH Terms: conditions — Phobia, Social | interventions — Behavior Therapy; Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exposure in vivo (Experimental): This treatment will consist of 10 sessions (twice a week) of exposure therapy based on the protocol used previously in exposure therapy for social anxiety disorder by Scholing & Emmelkamp (1993).
  Interventions: Behavioral: Exposure in vivo
- Virtual Reality Exposure Therapy (Experimental): This treatment consists of 10 sessions (twice a week) of exposure therapy by using virtual environments.
  The difference between the exposure in vivo and virtual reality exposure therapy is the exposure component, which will be delivered in vivo in one condition and through the Head Mounted Display (HMD) in the other condition.
  Interventions: Behavioral: Virtual Reality Exposure Therapy
- Wait-list (No Intervention): Participants on the wait-list will be offered either exposure in vivo or in virtual reality after a waiting period of five weeks.

INTERVENTIONS:
Behavioral: Exposure in vivo
  Other Names: Behavior Therapy
  Arms: Exposure in vivo
Behavioral: Virtual Reality Exposure Therapy
  Other Names: Virtual Reality Therapy
  Arms: Virtual Reality Exposure Therapy

SUMMARY:
The current study aims at comparing the efficacy of exposure in vivo and exposure via virtual reality for social anxiety disorder. 70 patients with social anxiety disorder will be randomized to either one of the active conditions or to a waiting-list condition. Participants on the waiting-list will be offered either exposure in vivo of in virtual reality after a waiting period of five weeks. Levels of psychopathology will be assessed at pre- and post-treatment as well as three and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old
* a primary diagnosis of social anxiety disorder as measured with the SCID
* fluency in Dutch.

Exclusion Criteria:

* psychotic episodes in the past, suicidal intentions or substance dependence.
* behavior therapy in the preceding one year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline: Liebowitz Social Anxiety Scale-Self report | Pre-treatment to post-treatment (5 weeks), three months follow-up, and 12 months follow-up.
  Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.
Change from baseline: Fear of Negative Evaluation Scale | Pre-treatment to post-treatment (5 weeks), three months follow-up, and 12 months follow-up.
  Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.

SECONDARY OUTCOMES:
Change from baseline: Behavioral Assessment Task (BAT), Public Speaking Performance Scale | Pre-treatment to post-treatment (5 weeks)
  The BAT consists of a videotaped 5 minute impromptu speech in front of two confederates. The Public Speaking Performance Scale will be used to evaluate the performance during the speech, both by patients and indipendent raters.
  Change from pre-treatment to post-treatment (5 weeks) will be examined.
Change from baseline: Structured Clinical Interview for DSM-IV (Social Phobia Module) | Pre-treatment to three months follow-up.
  Change in diagnosis of Social Phobia from pre-treatment to three months follow-up.
Change from baseline: Depression Anxiety Stress Scale | Pre-treatment to post-treatment (5 weeks), three months follow-up, 12 months follow-up.
  Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.
Change from baseline: Personality Disorder Belief Questionnaire | Pre-treatment to post-treatment (5 weeks), three months follow-up, 12 months follow-up.
  Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.
Change from baseline: Eurohis Quality of Life Scale | Pre-treatment to post-treatment (5 weeks), three months follow-up, 12 months follow-up.
  Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.

OTHER OUTCOMES:
Change from baseline and in-treatment change: Focus of Attention Questionnaire | Pre-treatment to post-treatment (5 weeks), change during the course of four weeks of exposure therapy (session 3 until 9)
  Focus of Attention will be assessed during the course of four weeks of exposure therapy that will take place twice a week (session 3 until 9). Change from pre-treatment to post-treatment (5 weeks) as well as change during treatment (four weeks) will be assessed.
In-treatment change: Social Phobia Weekly Summary Scale | Change from session to session during the course of five weeks (i.e., session 1 until 10)
  The Social Phobia Weekly Summary Scale will be used in each session during the course of the treatment that will take place twice a week (session 1 until 10). Change during treatment will be assessed.
Change from baseline:Social Cost Questionnaire | Pre-treatment to session 7 (3,5 weeks) and post-treatment (5 weeks)
  Change from pre-treatment to sessino 7 (3,5 weeks) and to post-treatment (5 weeks).
Experiences in Close Relationships Questionnaire | Pre-treatment
In treatment change: Self-efficacy for Social Situations | Change from session to session during the course of five weeks (i.e., session 1 until 10)
  Self-efficacy will be used in each session during the course the treatment that will take place twice a week (session 1 until 10). Change during treatment will be assessed (5 weeks).
In-treatment change: Working Alliance Inventory -Short Revised | Session 3 to session 6 (two weeks)
  Change during treatment (with an expected average of two weeks) will be assessed.
Simulator Sickness Questionnaire | Session 2 (first week of treatment)
  This scale will be used in the Virtual Reality condition only
Credibility and Expectancy Questionnaire | Session 3 (second week of treatment)
In-treatment change: Ingroup Presence Questionnaire | Session 2 to session 3 (one week) and session and 6 (three weeks).
  This scale will be used in the Virtual Reality condition only to measure change in the sense of presence from session 2 to session 3 (one week) and session 6 (three weeks).
Change from baseline: Dot-Probe Task | Pre-treatment to post-treatment (5 weeks), three months follow-up, and 12 months follow-up.
  An implicit measure to assess attentional bias in social phobia. Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.
Change from baseline: Approach Avoidance Task | Pre-treatment to post-treatment (5 weeks), three months follow-up, and 12 months follow-up.
  A computer task to assess automatic approach and avoidance tendencies by measuring reaction times for pushing away or pulling closer faces with a joystick. Change from pre-treatment to post-treatment (5 weeks), 3 months follow-up and 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul GM Emmelkamp, PhD, Principal Investigator — University of Amsterdam; Nexhmedin Morina, PhD, Study Director — University of Amsterdam
Locations (1):
- University of Amsterdam, Department of Clinical Psychology, Amsterdam, Netherlands

REFERENCES:
- [Derived] Kampmann IL, Emmelkamp PMG, Morina N. Cognitive predictors of treatment outcome for exposure therapy: do changes in self-efficacy, self-focused attention, and estimated social costs predict symptom improvement in social anxiety disorder? BMC Psychiatry. 2019 Feb 22;19(1):80. doi: 10.1186/s12888-019-2054-2. PMID 30795749